CLINICAL TRIAL: NCT05039710
Title: A Double-Blind, Placebo-Controlled, Randomized, Single Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneously Administered JNJ-75220795 in Japanese Participants
Brief Title: A Study of JNJ-75220795 in Japanese Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Judgement
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CR109081; 75220795NAS1002 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2021-09-01; First posted 2021-09-09 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Fatty Liver
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort 1: JNJ-75220795 or Placebo (Experimental): Participants will receive single subcutaneous (SC) dose of JNJ-75220795 Dose 1 or matching placebo on Day 1 in Cohort 1.
  Interventions: Drug: JNJ-75220795; Other: Placebo
- Cohort 2: JNJ-75220795 or Placebo (Experimental): Participants will receive single SC dose of JNJ-75220795 Dose 2 or matching placebo on Day 1 in Cohort 2.
  Interventions: Drug: JNJ-75220795; Other: Placebo

INTERVENTIONS:
Drug: JNJ-75220795 — JNJ-75220795 will be administered as SC injection.
Other: Placebo — Matching placebo will be administered as SC injection.

SUMMARY:
The purpose of this study is to assess the safety and tolerability of single subcutaneous (SC) dose of JNJ-75220795 in Japanese participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants with certain genetic predispositions to non-alcoholic fatty liver disease (NAFLD) determined at screening
* Presence of liver steatosis at screening
* Participants on anti-hypertensive and/or lipid lowering medications and/or glucose lowering medications must be on stable dose(s) for at least 4 weeks prior to screening
* Body mass index between 18 kilograms per meter square (kg/m^2) and 40 kg/m^2 inclusive, and body weight stable defined as no more than 5 percent (%) body weight loss or gain within 3 months prior to screening (based on participant's report) and no more than 5% body weight loss or gain from screening to randomization

Exclusion Criteria:

* Known allergies, hypersensitivity, or intolerance to excipients
* History of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-HCV) positive, or other clinically active liver disease, or tests positive for HbsAg or anti-HCV at screening. And/or history of human immunodeficiency virus (HIV) antibody positive, or tests positive for HIV or syphilis at screening
* Participants with clinical or biochemical (international normalized ratio [INR] greater than [>] 1.2, or platelet count less than [<] lower limits of normal [LLN]) evidence of hepatic decompensation at screening or baseline
* Estimated glomerular filtration rate (eGFR) by Japanese eGFR formula below 60 milliliters per minute [mL/min] at screening
* Thyroid stimulating hormone (TSH) levels, free triiodothyronine (FT3) and free thyroxine (FT4) outside normal limits of the clinical laboratory's reference range at screening

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-emergent Signs and Symptoms/Adverse Events (AEs) | Up to Day 168
  Number of participants with treatment-emergent signs and symptoms/adverse events (including allergic reactions/hypersensitivity and local injection site reactions) will be reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Treatment-emergent adverse events (TEAEs) are defined as AEs with onset or worsening on or after date of first dose of study treatment.
Number of Participants With Change From Baseline in Vital Signs Abnormalities | Baseline, Up to Day 168
  Number of participants with change from baseline in vital signs abnormalities including body temperature (axillary), pulse, respiratory rate and blood pressure will be reported.
Number of Participants With Change From Baseline in Clinical Laboratory Abnormalities | Baseline, Up to Day 168
  Number of participants with change from baseline in clinical laboratory abnormalities including hematology, serum chemistry and urinalysis will be reported.
Number of Participants With Change From Baseline in Physical Examination Abnormalities | Baseline, Up to Day 168
  Number of participants with change from baseline in physical examination abnormalities will be reported.
Number of Participants With Change From Baseline in Electrocardiogram (ECG) Abnormalities | Baseline, Up to Day 168
  Number of participants with change from baseline in ECG abnormalities will be reported.

SECONDARY OUTCOMES:
Percent Change in Liver Fat Content Measured by Magnetic Resonance Imaging - Proton Density Fat Fraction (MRI-PDFF) | From Baseline to Weeks 6, 12, 18, and 24
  Percent change in liver fat content as measured by MRI-PDFF will be reported.
Maximum Observed Plasma Concentration (Cmax) of JNJ-75220795 | Predose up to 48 hours postdose (up to Day 3)
  Cmax of JNJ-75220795 will be reported.
Time to Reach Maximum Observed Plasma Concentration (Tmax) of JNJ-75220795 | Predose up to 48 hours postdose (up to Day 3)
  Tmax of JNJ-75220795 will be reported.
Apparent Elimination Half-Life (t1/2) of JNJ-75220795 | Predose up to 48 hours postdose (up to Day 3)
  t1/2 is defined as apparent elimination half-life associated with the terminal slope of the semilogarithmic drug concentration-time curve.
Area Under the Plasma Concentration Time Curve of JNJ-75220795 from Time Zero to Infinite time (AUC [0-Infinity]) | Predose up to 48 hours postdose (up to Day 3)
  AUC (0-Infinity) is defined as the area under the plasma concentration versus time curve of JNJ-75220795 from time zero to infinite time.
Area Under the Plasma Concentration versus Time Curve of JNJ-75220795 from Time Zero to Time of the Last Measurable Concentration (AUC [0-Last]) | Predose up to 48 hours postdose (up to Day 3)
  AUC (0-Last) is defined as area under the plasma concentration versus time curve of JNJ-75220795 from time zero to time of the last measurable concentration.
Total Apparent Clearance (CL/F) of JNJ-75220795 | Predose up to 48 hours postdose (up to Day 3)
  CL/F is defined as total apparent clearance of JNJ-75220795.
Apparent Volume of Distribution (Vd/F) of JNJ-75220795 | Predose up to 48 hours postdose (up to Day 3)
  Vd/F is defined as apparent volume of distribution of JNJ-75220795.
Number of Participants with Treatment Emergent Anti-drug Antibody (ADA) | Up to Day 168
  Number of participants with treatment emergent ADA will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (4):
- Japan (4):
  - Souseikai Fukuoka Mirai Hospital, Fukuoka
  - Medical Corporation Heishinkai ToCROM Clinic, Shinjuku-ku
  - Heishinkai TOCROM Clinic, Suita
  - Sumida Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency